CLINICAL TRIAL: NCT06310473
Title: Efficacy and Safety of Neoadjuvant Cadonilimab and Chemotherapy for Locally Advanced Esophagogastric Junction and Gastric Cancer : a Prospective, Open-label, Single-Arm Phase II Study
Brief Title: Neoadjuvant Cadonilimab Plus Chemotherapy for Locally Advanced Esophagogastric Junction and Gastric Cancer Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2023-582
Record Dates: First submitted 2024-02-20; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer; Esophagogastric Junction Cancer
Keywords: bispecific antibody; Neoadjuvant; Immunotherapy and Chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab Plus Chemotherapy (Experimental): Neoadjuvant Immunotherapy and Chemotherapy：Cadonilimab+Oxaliplatin+Capecitabine, every 3 weeks for 3 cycles;
  Adjuvant chemotherapy： Oxaliplatin+Capecitabine, every 3 weeks for 3-5 cycles;
  Interventions: Drug: Cadonilimab; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Cadonilimab — 10mg/kg intravenous (IV) every 3 weeks ;
  Other Names: AK104
Drug: Oxaliplatin — 130mg/m², iv drip for 2h, d1, q3w;
Drug: Capecitabine — 1000mg/m² po, Bid, d1-14, q3w ;

SUMMARY:
For locally advanced esophagogastric junction and gastric cancer, neoadjuvant chemotherapy can downstage T and N stage,treated distant micrometastases early , and finally improve the long-term survival. Combination of perioperative PD-1 antibody and chemotherapy for locally advanced esophagogastric junction and gastric cancer could be a novel therapy to increase response rate and reduce recurrence rate.Cadonilimab, a tetravalent bispecific antibody targeting PD-1 and CTLA-4, is designed to retain the efficacy benefit of combination of PD-1 and CTLA-4 and improve on the safety profile of the combination therapy. The aim of this study is to evaluate the efficacy and safety of cadonilimab Plus Chemotherapy for Locally Advanced Esophagogastric Junction and Gastric Cancer.

DETAILED DESCRIPTION:
Locally advanced esophagogastric junction and gastric cancer could be cured by multi-disciplinary therapies including surgery, chemotherapy and radiotherapy. Neoadjuvant chemotherapy can downstage T and N stage, treated distant micrometastases early before local therapy has begun, and finally improve the long-term survival. However, the therapeutic effects remain unsatisfactory.Cadonilimab (AK104), a novel bispecific antibody simultaneously targeting PD-1 and CTLA-4, was designed to boost anti-tumor activity with a favorable safety profile.This study was a single arm, open-label clinical study to evaluate the efficacy and safety of combination with Cadonilimab and Chemotherapy for neoadjuvant treatment of resectable locally advanced adenocarcinoma of the gastro-esophageal junction.

ELIGIBILITY:
Key Inclusion Criteria:

1. Confirmed gastric and gastroesophageal junction adenocarcinoma by Gastroscopic biopsy histopathological examination.
2. Imaging (CT/MRI) and diagnostic laparoscopy confirmed at the stage of cT3-4aN1-3M0(AJCC 8th) .
3. Physical condition and organ function allow for for larger abdominal surgery.
4. Adequate haematological, renal and liver function.

Key Exclusion Criteria:

1. Patients who have HER2 positive confiemed with IHC3+ or IHC2+ and FISH positive.
2. Confirmed at stage IV (AJCC 8th) or unresectable by investigator.
3. Prior chemotherapy, radiotherapy, surgery immunotherapy or molecular targeted therapy for gastric cancer.
4. Patients are allergic to study medication and its ingredients.
5. Known active autoimmune diseases.
6. Presence of other uncontrolled serious medical conditions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete remission rate (pCR) | up to 1 years
  Pathological complete response (pCR) rate is defined as the proportion of participants whose tumor in the stomach and lymph node completely disappeared, as determined by a pathologist.

SECONDARY OUTCOMES:
Major pathologic response，MPR | up to 1 years
  Major pathological response (MPR) rate is defined as the proportion of participants whose percentage of residual tumor in the stomach and lymph node decreased to < 10%, as determined by a pathologist
R0 resection rate | up to 1 years
  Rate of microscopically margin-negative resection
Objective Response Rate (ORR) | up to 3 years
  defined as the percentage of participants who achieve a best overall response of complete response or partial response assessed according to mRECIST v1.1 for assessment of response in malignant pleural mesothelioma.
Disease Control Rate (DCR) | up to 3 years
  defined as the percentage of participants who achieve a best overall response of complete response, partial response, or stable disease assessed according to mRECIST v1.1 for assessment of response in malignant pleural mesothelioma.
3-year disease-free survival rate of 3year (DFS) | up to 3 years
  3 years disease-free survival (DFS) rate is defined as proportion of participants who have no recurrence or metastasis after 3 years of radical treatment
Overall Survival (OS) | up to 3 years
  defined as the time between the date of first dose of study drug and the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Guoxin Li, M.D., Ph.D, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No